CLINICAL TRIAL: NCT00793403
Title: Current Adoption Of Composite Indices In Evaluating Rheumatoid Arthritis Patients: An Observational Study ("NEW INDICES Study")
Brief Title: Current Adoption of Composite Indices in Evaluating Rheumatoid Arthritis Patients: An Observational Study
Acronym: New Indices
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A1-102317; 0881A-102317 ; B1801118
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2012-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Observational cohort; prospectives; multicentre; the Italian study RA patient CLARA and PRO-CLARA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: As per routine clinical care
  Interventions: Other: As per routinary clinical care

INTERVENTIONS:
Other: As per routinary clinical care — As per routine clinical care
  Other Names: Observational study

SUMMARY:
This is an observational study of composite indices, including the CLARA (CLinical ARthritis Activity) index, in rheumatoid arthritis (RA) patients in routine clinical practice in Italy in order to evaluate clinical remission and low disease activity. Data will be collected only from patients providing informed consent. In this study we aimed to assess the psychometric properties of a new composite instrument termed CLinical ARthritis Activity (PRO-CLARA) that uses only three PRO measures from among the 7 ACR Core Data Set. We hypothesized that this index would facilitate rapid and easy RA activity assessment in daily routine.

DETAILED DESCRIPTION:
All patients who respond to inclusion/exclusion criteria at baseline will be considered valuable for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older with diagnosis of RA based on the 1987 American College of Rheumatology (ACR) criteria and in accordance with local guidelines.
* Patients eligible to anti-TNF therapy
* Patients naïve to anti-TNFa drugs
* Patients with radiography (hands and feet) executed by 6 months before the baseline or at baseline according to modified Sharp Van der Hejde method [Sharp JT et al. 1985; Sharp JT. Et al. 1989; Van der Heijde DM et al. 1989] Patients capable of understanding and completing the questionnaire Patients capable of understanding and signing an informed consent form

Exclusion Criteria:

* Patients with tumors
* Patients already included in clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Torino, Italy

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A1-102317&StudyName=Current%20adoption%20of%20composite%20indices%20in%20evaluating%20rheumatoid%20arthritis%20patients%3A%20An%20Observational%20Study

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Active Rheumatoid Arthritis (RA) participants who were partial or non-responders to the previous Disease Modifying Anti Rheumatic Drugs (DMARDs) treatment were prescribed with anti-Tumor Necrosis Factor (TNF) therapy (infliximab, etanercept, and adalimumab) as per usual clinical practice and observed for 12 months.
Period: Overall Study
Arm/Group | All Participants
Started | 293
Completed | 220
Not Completed | 73
Not completed — Other | 73

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 220
Age Continuous [Mean (Standard Deviation); unit: Years] | 55.65 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Remission as Per Modified American College of Rheumatology (Modified ACR) Criteria at Month 6
Description: Modified ACR: participant considered in RA remission if at any time point 1) participant satisfied all of the following criteria: tender joint count(TJC) less than or equal to(<=)1;swollen joint count(SJC)<=1 (TJC, SJC based on 28-joints);C-reactive protein(CRP)<=1 milligram/deciliter(mg/dL); patient global assessment (PtGA) <=1 (assessed on 0-10 centimeter[cm] visual analog scale[VAS]) or 2) participant had Simplified Disease Activity Index score of <=3.3 (SDAI, numerical sum of 5 outcome parameters: TJC, SJC, PtGA, physician global assessment [PGA, assessed on 0-10 cm VAS], and CRP [mg/dL]).
Time Frame: Month 6
Population: Data was not analyzed as per planned analysis because it was not considered significant to assess the outcome according to clinical opinion.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Primary Outcome: Percentage of Participants With Remission as Per Modified American College of Rheumatology (Modified ACR) Criteria at Month 12
Description: Modified ACR: participant was considered in RA remission if at any time point 1) participant satisfied all of the following criteria: TJC <=1; SJC <=1 (TJC, SJC based on 28-joints); CRP <=1 mg/dL; PtGA<=1 (assessed on 0-10 centimeter[cm] visual analog scale[VAS]) or 2) participant had SDAI score of <=3.3 (SDAI: the numerical sum of 5 outcome parameters: TJC, SJC, PtGA, PGA [assessed on 0-10 cm VAS], and CRP [mg/dL]).
Time Frame: Month 12
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Primary Outcome: Minimal Disease Activity: Outcome Measures in Rheumatology Arthritis Clinical Trials (OMERACT) at Month 6
Description: OMERACT minimal disease activity: participant considered with minimal disease activity if he/she met 5 of 7 criteria: Pain <=2 (assessed on a 0-10 cm VAS, 0 cm=no pain and 10 cm=worst possible pain); SJC <=1; TJC <=1 (SJC, TJC based on 28-joints); Health Assessment Questionnaire (HAQ) <=0.5 (assessment of ability to perform task on 0-3 point scale, 0=least difficulty and 3=extreme difficulty); PGA <=1.5; PtGA <=2 (PGA, PtGA: assessed on 0-10 cm VAS, higher score = greater affection due to disease activity); erythrocyte sedimentation rate (ESR) <=20 millimeter per hour (mm/hr).
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Primary Outcome: Minimal Disease Activity: Outcome Measures in Rheumatology Arthritis Clinical Trials (OMERACT) at Month 12
Description: OMERACT minimal disease activity: participant considered with minimal disease activity if he/she met 5 of 7 criteria: Pain <=2 (assessed on a 0-10 cm VAS, 0 cm=no pain and 10 cm=worst possible pain); SJC <=1; TJC <=1 (SJC, TJC based on 28-joints); HAQ <=0.5 (assessment of ability to perform task on 0-3 point scale, 0=least difficulty and 3=extreme difficulty); PGA <=1.5; PtGA <=2 (PGA, PtGA: assessed on 0-10 cm VAS, higher score = greater affection due to disease activity); ESR <=20 mm/hr.
Time Frame: Month 12
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

5. Primary Outcome: Minimal Disease Activity: Italian Group for the Study of Early Arthritis (GISEA) at Month 6
Description: GISEA minimal disease activity criteria: a participant was considered with minimal disease activity if he/she met the following criteria: SJC <=2 (based on 28-joints); HAQ <=0.5 (assessment of ability to perform task on 0-3 point scale, 0=least difficulty and 3=extreme difficulty); and ESR <=20 mm/hr.
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

6. Primary Outcome: Minimal Disease Activity: Italian Group for the Study of Early Arthritis (GISEA) at Month 12
Description: as for outcome 5
Time Frame: Month 12
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

7. Primary Outcome: Number of Swollen Joints (SJC) and Tender Joints (TJC) at Month 6
Description: Number of swollen joints was determined by examination of 28 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1.
  Number of tender joints was determined by examining 28 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1.
Time Frame: Month 6
Population: Analysis population included all participants who were enrolled in the study. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | All Participants
Number analyzed (Participants) | 217
Joints
  SJC | 2.80 (3.84)
  TJC | 4.62 (5.01)

8. Primary Outcome: Number of Swollen Joints (SJC) and Tender Joints (TJC) at Month 12
Description: as for outcome 7
Time Frame: Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | All Participants
Number analyzed (Participants) | 155
Joints
  SJC | 1.28 (2.72)
  TJC | 2.35 (3.47)

9. Primary Outcome: Disease Activity Score Based on 28-joints Count (DAS28) at Month 6
Description: DAS28 calculated from SJC and TJC using the 28 joints count, the ESR (mm/hr) and PtGA of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10 cm VAS; higher scores indicated greater affectation due to disease activity). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28 <= 3.2 implied low disease activity and > 3.2 to 5.1 implied moderate to high disease activity, and DAS28 < 2.6 = remission.
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

10. Primary Outcome: Disease Activity Score Based on 28-joints Count (DAS28) at Month 12
Description: as for outcome 9
Time Frame: Month 12
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

11. Primary Outcome: Simplified Disease Activity Index (SDAI) at Month 6
Description: The SDAI is the numerical sum of five outcome parameters: TJC and SJC (based on a 28-joint assessment), PtGA and PGA (assessed on 0-10 cm VAS; higher scores=greater affection due to disease activity), and CRP (mg/dL). SDAI total score= 0-86. SDAI <=3.3 indicates disease remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high disease activity.
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

12. Primary Outcome: Simplified Disease Activity Index (SDAI) at Month 12
Description: as for outcome 11
Time Frame: Month 12
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

13. Primary Outcome: Rheumatoid Arthritis Disease Activity Index (RADAI) at Month 6
Description: RADAI:self-assessed measure of disease activity in RA. Consists of 5 items: global disease activity(GDA) in past 6 months; current disease activity(CDA) as measured by SJC and TJC; current arthritis pain; current duration of morning stiffness; current TJC. GDA,CDA and pain were scored on an 11-point numerical rating scale,0=no disease activity/pain to 10=extreme disease activity/pain. Current morning stiffness and TJC were transformed to a 0-10 point scale,higher scores=more disease activity. RADAI total score=sum of individual items divided by 5;range 0-10, higher score=more disease activity.
Time Frame: Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 217
Units on a scale | 3.26 (1.78)

14. Primary Outcome: Rheumatoid Arthritis Disease Activity Index (RADAI) at Month 12
Description: RADAI:self-assessed measure of disease activity in RA. Consists of 5 items: GDA in past 6 months; CDA as measured by SJC and TJC; current arthritis pain; current duration of morning stiffness; current TJC. GDA,CDA and pain were scored on an 11-point numerical rating scale,0=no disease activity/pain to 10=extreme disease activity/pain. Current morning stiffness and TJC were transformed to a 0-10 point scale,higher scores=more disease activity. RADAI total score=sum of individual items divided by 5;range 0-10, higher score=more disease activity.
Time Frame: Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 137
Units on a scale | 2.83 (1.89)

15. Primary Outcome: Clinical Disease Activity Index (CDAI) at Month 6
Description: The CDAI is the numerical sum of 4 outcome parameters: TJC and SJC (based on a 28-joint assessment), PtGA and PGA (assessed on 0-10 cm VAS; higher scores=greater affection due to disease activity). CDAI total score = 0-76. CDAI <= 2.8 indicates disease remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high disease activity.
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

16. Primary Outcome: Clinical Disease Activity Index (CDAI) at Month 12
Description: as for outcome 15
Time Frame: Month 12
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

17. Primary Outcome: Patient Reported Outcomes - Clinical Arthritis Activity (PRO-CLARA ) at Month 6
Description: PRO-CLARA:self-administered index of RA activity. Consists of 3-items: participant's physical function (12 questions each scored on a 0 [without any difficulty] to 4 [unable to do] point scale); TJC(based on 16-joints, tenderness assessed on 0 [none] to 3 [severe] point scale); PtGA (participant rated disease activity on 0-10 cm VAS, 0=very well, 10 cm=very poorly). Participant's physical function and TJC were transformed on a 0-10 point scale, higher scores=more disease activity. PRO-CLARA total score=sum of scores of all 3 items divided by 3, range= 0-10, higher scores=more disease activity.
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

18. Primary Outcome: Patient Reported Outcomes - Clinical Arthritis Activity (PRO-CLARA ) at Month 12
Description: as for outcome 17
Time Frame: Month 12
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

19. Primary Outcome: Clinical Arthritis Activity (CLARA) Index at Month 6
Description: CLARA: index of RA activity. Consists of 3-items: participant's physical function (12 questions each scored on a 0 [without any difficulty] to 4 [unable to do] point scale); TJC (based on 16-joints, tenderness assessed on 0 [none] to 3 [severe] point scale); SJC (based on 28-joints). Each item was transformed on a 0-10 point scale, higher scores=more disease activity. CLARA total score=sum of scores of all 3 items divided by 3, range= 0-10, higher scores=more disease activity.
Time Frame: Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 215
Units on a scale | 1.79 (1.37)

20. Primary Outcome: Clinical Arthritis Activity (CLARA) Index at Month 12
Description: as for outcome 19
Time Frame: Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 137
Units on a scale | 1.39 (1.33)

21. Primary Outcome: Patient Global Assessment (PtGA) of Disease Activity at Month 6
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 10 cm VAS, where 0 cm = very well and 10 cm = very poorly.
Time Frame: Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | All Participants
Number analyzed (Participants) | 219
cm | 3.71 (2.23)

22. Primary Outcome: Patient Global Assessment (PtGA) of Disease Activity at Month 12
Description: as for outcome 21
Time Frame: Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | All Participants
Number analyzed (Participants) | 143
cm | 3.35 (2.21)

23. Primary Outcome: Physician Global Assessment (PGA) of Disease Activity at Month 6
Description: Physician Global Assessment of Arthritis was measured on a 0 to 10 cm VAS, where 0 cm = very good and 10 cm = very bad.
Time Frame: Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | All Participants
Number analyzed (Participants) | 219
cm | 3.11 (2.04)

24. Primary Outcome: Physician Global Assessment (PGA) of Disease Activity at Month 12
Description: Physician Global Assessment of Arthritis was measured on a 0 to 10 cm VAS, where 0 cm = very good and 10 cm = very bad.
Time Frame: Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | All Participants
Number analyzed (Participants) | 147
cm | 2.60 (1.95)

25. Primary Outcome: Visual Analog Fatigue Scale (VAFS) at Month 6
Description: Participants assessed their fatigue using a 0 - 100 mm VAS, where 0 mm = no fatigue and 100 mm = worst possible fatigue.
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

26. Primary Outcome: Visual Analog Fatigue Scale (VAFS) at Month 12
Description: Participants assessed their fatigue using a 0 - 100 mm VAS, where 0 mm = no fatigue and 100 mm = worst possible fatigue.
Time Frame: Month 12
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

27. Primary Outcome: C-reactive Protein (CRP) at Month 6
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. Normal range of CRP is <1 mg/dL. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 184
mg/dL | 2.16 (4.07)

28. Primary Outcome: C-reactive Protein (CRP) at Month 12
Description: as for outcome 27
Time Frame: Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 136
mg/dL | 1.63 (2.25)

29. Primary Outcome: Erythrocyte Sedimentation Rate (ESR) at Month 6
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 mm/hr. A higher rate is consistent with inflammation.
Time Frame: Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | All Participants
Number analyzed (Participants) | 200
mm/hr | 26.02 (19.19)

30. Primary Outcome: Erythrocyte Sedimentation Rate (ESR) at Month 12
Description: as for outcome 29
Time Frame: Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | All Participants
Number analyzed (Participants) | 152
mm/hour | 21.92 (15.65)

31. Primary Outcome: Number of Participants With Rheumatoid Factor (RF) at Month 6
Description: RF is the auto antibody directed against immunoglobulin G (IgG) and its concentration is observed in human serum or plasma. RF value higher than 20 units per milliliter (U/mL) is considered positive.
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

32. Primary Outcome: Number of Participants With Rheumatoid Factor (RF) at Month 12
Description: RF is the auto antibody directed against immunoglobulin G (IgG) and its concentration is observed in human serum or plasma. RF value higher than 20 U/mL is considered positive.
Time Frame: Month 12
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

33. Primary Outcome: Patient's General Health Assessment at Month 6
Description: Participants answered: "How would you describe your general health today?" Participants assessed their general health using a 0 - 10 cm VAS, where 0 cm = very well and 10 cm = very poor.
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

34. Primary Outcome: Patient's General Health Assessment at Month 12
Description: as for outcome 33
Time Frame: Month 12
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

35. Primary Outcome: Patient Assessment of Arthritis Pain at Month 6
Description: Participants rated the severity of arthritis pain on a 0 to 10 cm VAS, where 0 cm = no pain and 10 cm = most severe pain.
Time Frame: Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | All Participants
Number analyzed (Participants) | 219
cm | 3.58 (2.31)

36. Primary Outcome: Patient Assessment of Arthritis Pain at Month 12
Description: as for outcome 35
Time Frame: Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | All Participants
Number analyzed (Participants) | 143
cm | 3.29 (2.31)

37. Primary Outcome: Duration of Morning Stiffness at Month 6
Description: Duration of morning stiffness: Time elapsed when participant woke up in morning and was able to resume normal activities without stiffness in minutes. Increase in stiffness duration from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

38. Primary Outcome: Duration of Morning Stiffness at Month 12
Description: as for outcome 37
Time Frame: Month 12
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

39. Primary Outcome: Health Assessment Questionnaire (HAQ) at Month 6
Description: HAQ: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 218
Units on a scale | 0.83 (0.65)

40. Primary Outcome: Health Assessment Questionnaire (HAQ) at Month 12
Description: as for outcome 39
Time Frame: Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 139
Units on a scale | 0.68 (0.66)

41. Primary Outcome: Recent-Onset Arthritis Disability (ROAD) at Month 6
Description: ROAD questionnaire: valid and responsive tool for measuring functional ability in RA participants. Consists of 12-items related to fine movements of upper extremity, locomotor activities of lower extremity, and activities that involve both upper and lower extremities. For each item participant rated the level of difficulty over the past week on a 5-point scale ranging from 0 (without any difficulty) to 4 (unable to do). Total ROAD score were transformed to a 0 to 10 point scale, where 0 = best status and 10 = poorest status.
Time Frame: Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 218
Units on a scale | 2.28 (1.88)

42. Primary Outcome: Recent-Onset Arthritis Disability (ROAD) at Month 12
Description: as for outcome 41
Time Frame: Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 138
Units on a scale | 1.97 (1.92)

43. Primary Outcome: Radiological Assessment of Hands and Feet Based on Sharp-van Der Hejde (SvH) Scoring Method at Month 6
Description: SvH method included 16 areas for erosions and 15 areas for joint space narrowing (JSN) and subluxation/luxation in each hand, 6 areas for erosions and 6 areas for JSN and subluxation/luxation in each foot. Erosion per joint scored on 0-5 point scale; 0=normal joint to 5=complete collapse. Total erosion score for hands:0-160, for feet:0-120. JSN and subluxation/luxation scored on 0-4 point scale; 0=normal joint to 4= a bony ankylosis/a complete luxation of joint. Total JSN and subluxation/luxation score for hands:0-120, for feet:0-48. Total SvH score = 0-448; higher score=more erosion and JSN.
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

44. Primary Outcome: Radiological Assessment of Hands and Feet Based on Sharp-Van Der Hejde (SvH) Scoring Method at Month 12
Description: SvH method included 16 areas for erosions and 15 areas for JSN and subluxation/luxation in each hand, 6 areas for erosions and 6 areas for JSN and subluxation/luxation in each foot. Erosion per joint scored on 0-5 point scale; 0=normal joint to 5=complete collapse. Total erosion score for hands:0-160, for feet:0-120. JSN and subluxation/luxation scored on 0-4 point scale; 0=normal joint to 4= a bony ankylosis/a complete luxation of joint. Total JSN and subluxation/luxation score for hands:0-120, for feet:0-48. Total SvH score = 0-448; higher score=more erosion and JSN.
Time Frame: Month 12
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 4/293
Other Adverse Events (participants affected / at risk) | 7/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=293)
Hospitalization for dermatitis (General disorders) | 1
Local aedematous reaction, hard and pain (General disorders) | 1
Suspect of feocromocitoma (General disorders) | 1
(General disorders) | 1 — Information was collected from phone log data and no information was available about serious event occurred.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=293)
Skin rash on abdomen and chest (General disorders) | 1
Foot finger infection (General disorders) | 1
Visus disorder (General disorders) | 1
Erythematous reaction in the injection site (General disorders) | 1
Vasculite episode (General disorders) | 1
Defluvium Capillorum (General disorders) | 1
Cystitis with fever (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.